CLINICAL TRIAL: NCT07147842
Title: Rutin Therapy Reduces Ulcerative Colitis Disease Activity By Inhibiting The NOD-Like Receptor Protein 3 (NLRP3) Inflammasome: A Molecular Assessment in a Case-Control Study
Brief Title: Rutin Therapy Role in Reducing Ulcerative Colitis Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Afnan El Gindy, Lecturer of Physiology, Faculty of Medicine, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC 3.7.2025
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Rutin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ulcerative Colitis-A (UC-A) (Active Comparator): Patients diagnosed with active Ulcerative Colitis were assigned as group UC-A
  Interventions: Drug: Rutin 500 MG; Diagnostic Test: fecal calprotectin
- Ulcerative Colitis-B (UC-B) (Active Comparator): Patients diagnosed with remission Ulcerative Colitis were assigned as control group UC-B
  Interventions: Other: Placebo; Diagnostic Test: fecal calprotectin
- Healthy Group (C) (Active Comparator): Healthy volunteers provided samples as negative controls; and was assigned as group C
  Interventions: Diagnostic Test: fecal calprotectin

INTERVENTIONS:
Drug: Rutin 500 MG — Rutin 500 mg capsules twice daily for 30 days
  Arms: Ulcerative Colitis-A (UC-A)
Other: Placebo — Placebo Tablets
  Arms: Ulcerative Colitis-B (UC-B)
Diagnostic Test: fecal calprotectin — Fecal calprotectin level was measured using an ELISA kit .

SUMMARY:
Ulcerative colitis (UC) is an inflammatory bowel disease characterized by oxidative stress and recurring inflammation in the colon. The condition can become chronic, spread, and lead to other complications.

A key player in the inflammation process is the NLRP3 inflammasome. This inflammasome's expression is heightened and activated by reactive oxygen species (ROS). Its activity is influenced by various factors, including the ubiquitin system, ion channels, and gut microbiota.

Rutin, a compound found in many fruits and vegetables, has been shown to have properties that help scavenge free radicals.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms suggestive of IBD;
* Patients with positive microscopic mucosal changes consistent with UC.

Exclusion Criteria:

* Patients with the presence of recurrent ulceration after surgical treatment, malignancy, or autoimmune disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Success Rate of Treatment Regimens in improving the ulcerative colitis. | 3~4 Months
  The proportion of patients who achieved a Simple Clinical Colitis Activity Index (SCCAI) score of 5 or less at the end of the study, which reflects the effectiveness of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt